CLINICAL TRIAL: NCT06117748
Title: Comparative Study Between the Effect of Volume-Controlled Ventilation and Pressure-Controlled Ventilation Volume Guaranteed in Obese Patients in Laparoscopic Assisted Surgery
Brief Title: Volume-Controlled Ventilation and Pressure-Controlled Ventilation Volume Guaranteed in Obese Patients in Laparoscopic-Assisted Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maamoun Maamoun Soliman, Assistant lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD 280 / 2022
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Volume-Controlled Ventilation; Pressure-Controlled Ventilation Volume Guaranteed; Obese; Laparoscopy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (PCV-VG): Pressure controlled ventilation-volume guaranteed (Experimental): Patients will receive pressure controlled ventilation-volume guaranteed
  Interventions: Other: Pressure controlled ventilation-volume guaranteed
- Group (VCV): Volume controlled ventilation (Other): Patients will receive Volume controlled ventilation
  Interventions: Other: Volume controlled ventilation

INTERVENTIONS:
Other: Pressure controlled ventilation-volume guaranteed — Respiratory parameters will be set as: actual tidal volume 8 mL/kg actual body weight, respiratory rate 12 breaths/min, PEEP of five mmHg, oxygen flow 1 L/min, fraction inspired oxygen (FiO2) 0.6, and I:E ratio of 1:2.
  Respiratory parameters will be kept constant if ETCO2 is <45 mmHg. When ETCO2 exceed 45 mmHg, respiratory rate or tidal volume will be adjusted to maintain ETCO2 below 45 mmHg.
  Arms: Group (PCV-VG): Pressure controlled ventilation-volume guaranteed
Other: Volume controlled ventilation — Respiratory parameters will be set as: actual tidal volume 8 mL/kg actual body weight, respiratory rate 12 breaths/min, PEEP of five mmHg, oxygen flow 1 L/min, fraction inspired oxygen (FiO2) 0.6, and I:E ratio of 1:2.
  Respiratory parameters will be kept constant if ETCO2 is <45 mmHg. When ETCO2 exceed 45 mmHg, respiratory rate or tidal volume will be adjusted to maintain ETCO2 below 45 mmHg.
  Arms: Group (VCV): Volume controlled ventilation

SUMMARY:
The aim of this study is to compare the efficacy of the pressure controlled ventilation volume-guaranteed (PCV-VG) versus volume-controlled ventilation (VCV) modes as regards lung compliance and oxygenation index in obese patients undergoing laparoscopic assisted surgery especially in Trendelenburg position.

DETAILED DESCRIPTION:
Obesity, defined as a Body Mass Index (BMI) >30 kg.m-2", is characterized by increased airway resistance, labored breathing and decreased respiratory system compliance. An increased rate of obese patients undergoing laparoscopic assisted surgery (LAS) is a health care concern due to anesthesia and ventilation difficulties in the obese population. Therefore, understanding the physiology and pathophysiology of lung function is an important issue during long-lasting LAS.

Carbon dioxide pneumoperitoneum with steep Trendelenburg positioning leads to a cranial displacement of the diaphragm and an increased volume of atelectasis, with a consequent decrease of total lung volume, lung compliance, and functional residual capacity. Thus, alleviation of increased airway pressure, improvement in oxygenation and CO2 elimination are the main goals during anesthetic management in laparoscopic assisted surgery.

In pressure controlled ventilation volume-guaranteed (PCV-VG) mode, the ventilator regulates the Peak Inspiratory Pressure (PIP) to achieve the optimal TV. To achieve the target volume, ventilator parameters are regularly changed without adjusting airway pressures. Hence, PCV-VG has the advantages of both Volume-Controlled Ventilation (VCV) and pressure controlled ventilation (PCV) to preserve the target minute ventilation while maintaining a low incidence of barotraumas.

PCV-VG is a type-controlled ventilation mode with a dual character as it has the criteria of both PCV and VCV. This recent ventilation mode which is one of the pressure regulated volume controlled (PRVC) that include Auto Flow ventilation, offers the ability to reduce the inspiratory pressure and as a result the incidence of barotrauma

ELIGIBILITY:
Inclusion Criteria:

1. Age: 16 - 60 years old.
2. Sex: both males and females.
3. Undergoing elective Laparoscopic Surgery.
4. Obese patient with Body Mass Index between ≥30 Kg/m2.
5. American society of Anesthesiologist (ASA) class I/ II.

Exclusion Criteria:

1. Patient refusal.
2. American society of Anesthesiology (ASA) III or IV.
3. Intraoperative hemodynamic instability.
4. Patients with pulmonary hypertension.
5. Obese patients on home O2 therapy
6. Pneumoperitoneum with CO2 with intra-abdominal pressure exceeding 15mmHg.
7. Anti-Trendelenburg position.
8. Asthmatic Patients.
9. Patients with advanced liver disease.
10. Patients with advanced renal disease.
11. Patients with advanced malignancy.
12. Pregnant females.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Oxygenation index | Till the end of surgery
  Oxygenation index =mean airway pressure × fraction of inspired oxygen (FiO2) × 100÷ Partial pressure of oxygen (PaO2)

SECONDARY OUTCOMES:
Mean arterial blood pressure | Till the end of surgery
  Mean arterial blood pressure (MAP) will be monitored 10 minutes before anesthesia induction , immediately before onset of pneumoperitoneum, every 10 minutes in the first hour, and at the end of surgery.
Heart rate | Till the end of surgery
  Heart rate (HR) will be monitored 10 minutes before anesthesia induction , immediately before onset of pneumoperitoneum, every 10 minutes in the first hour, and at the end of surgery.
Oxygen saturation SpO2 | Till the end of surgery
  Oxygen saturation SpO2 will be monitored 10 minutes before anesthesia induction , immediately before onset of pneumoperitoneum, every 10 minutes in the first hour, and at the end of surgery.
Arterial PCo2 | Till the end of surgery
  Arterial blood gases will be analyzed using a blood gas analyzer before anesthesia induction and every 10 minutes in the first hour for arterial oxygen tension (paO2) , arterial CO2 tension (paCO2).
Lung compliance | Till the end of surgery
  Lung mechanics readings included peak air way pressure (Ppeak), plateau pressure (Pplat), mean airway pressure (Pmean), dynamic and static compliance of the respiratory system will be recorded after intubation and every 10 minutes in the first hour

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.